CLINICAL TRIAL: NCT03597152
Title: Nutritional Supplementation for Extending Time Between Recurrent Urinary Tract Infections in Women: a Randomized Double Blind Cross-over Trial
Brief Title: Nutritional Supplementation for Recurrent Urinary Tract Infections in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AmPurity Nutraceuticals, LLC (Industry)
Collaborators: Arkansas Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMARU 001
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: uncomplicated recurrent urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): WelTract
  Interventions: Dietary Supplement: WelTract
- Control (Placebo Comparator): Inert Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: WelTract — Supplement commercially available from the sponsor containing powdered extracts from Hibiscus flowers and cranberry fruit, lactoferrin, D-mannose, and vitamins C and D
  Arms: Treatment
Dietary Supplement: Placebo — Inert placebo custom manufactured for the sponsor
  Arms: Control

SUMMARY:
The study will test the ability of specially formulated nutritional supplement capsules to extend the time between recurrent urinary tract infections in women. This objective will be completed by enrolling women who have suffered from 3-4 uncomplicated UTIs in the past 12 months into a double blind placebo controlled cross-over trial. Cross-over and study completion are triggered by the next two UTI recurrences. The goal of the study is for the supplement to extend the time to the next UTI for study participants as compared to placebo.

DETAILED DESCRIPTION:
Background: Recurrent urinary tract infections (UTIs), i.e. having three or more infections in 12 months, present a common and serious health problem for women. Long-term prophylactic antibiotic use is one treatment approach though there are currently no consensus treatment strategies for chronic recurrent UTIs which makes development of antibiotic resistant bacterial strains a major concern. Alternatively, nutritional supplements such as those based on cranberry and the sugar d-mannose, have shown some mixed success as a complementary treatment for UTIs. Thus, identification of a multi-ingredient nutritional supplement which could reduce the recurrence of UTIs when applied in conjunction with standard of care would be valuable to the heath and healthcare of women.

Objective: The study will test the efficacy of a twice-daily nutritional supplement for extending the time between recurrent UTIs in women. The supplement is a commercially available product (WelTract, AmPurity LLC) whose capsules contain extracts from Hibiscus flowers and cranberry fruit, lactoferrin, D-mannose, and vitamins C and D.

Methods: The study design will be a randomized double-blind placebo-controlled cross-over trial. The primary outcome will be time to recurrence of next UTI. Women (age 18-75 yrs) will be enrolled at a private urology clinic upon presentation of their 3rd or 4th simple cystitis of the lower urinary tract in the past 12 months. Randomization and product consumption will occur concurrently with standard of care treatment (acute antibiotics) of the infection. Resolution of the infection will be confirmed by urine culture and supplement or placebo consumption will continue until UTI recurrence which will trigger cross-over. Again, standard of care will ensue and consumption of the supplement or placebo will continue until UTI recurrence which triggers participant study completion. Cross-over is not forced and the maximum allowable time to cross-over and/or complete the study is one year per participant. Side-effects will be monitored and reported.

Analysis Plan: The study plans to enroll a maximum of 250 women, intending to ensure that 150 women complete the study. Statistical analysis will be performed using both the non-parametric Log Rank test and the Gail and Simon method, each with different primary outputs (statistical significance and effect size, respectively). Both of these methods are suitable for comparing paired time-to-event measures as found in a cross-over design. The baseline sample size (N=150) was calculated using the Cox Proportional Hazard method, at 85% desired power, an alpha level 0.05, a representative hazard ratio of 0.7 from prior cranberry treatment trials, and allowing for up to 40% of the subjects to not complete the study due to reasons such as withdrawal or dropout.

Clinical Significance: The daily consumption of a scientifically-based multi-ingredient nutritional supplement may provide a safe and practical means to extend the time until recurrence of the next UTI for women who have suffered 3-4 UTIs in the past 12 months when applied in combination with standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with symptoms of UTI
* Presentation of 3rd or 4th simple cystitis of lower tract in the past 12 months
* Active infection at enrollment, confirmed and documented in medical record
* Cognitive capacity to consent and ability to undergo the consent process in English

Exclusion Criteria:

* Known allergy or intolerance to supplement ingredients
* Pregnant or planning to become pregnant or lactating
* Unwilling to commit to birth control use
* Use of related nutritional supplements
* Unwilling to halt berry extracts, polyphenols, antioxidants, d-mannose, vitamins
* Taken WelTract in past six months
* Unwilling to avoid probiotics, yogurt, apple or cranberry juice, hibiscus tea
* Certain comorbid or physical conditions
* History of febrile UTI
* Bladder catheter or urethral stents
* Use of topical hormones in urogenital areas
* Diabetes (i.e. taking diabetic medications) or glycosuria
* Intestinal diseases with malabsorption (e.g. Crohn's and celiac diseases)
* Severe renal impairment or kidney stones
* Neural problems (spinal cord injury or Multiple Sclerosis)
* Immunocompromised individuals
* Rheumatoid arthritis
* Lupus
* HIV
* Taking steroids or immunobiologic medications
* Prophylactic antibiotic use (e.g. post-coital)
* Other physician judgement

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Not based on self-representation
Enrollment: 250 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-01-14 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
UTI Recurrence | Variable for each participant over course of up to one year
  Time to recurrence of next UTI

CONTACTS AND LOCATIONS:
Overall Officials: Richard D'Anna, MD, Principal Investigator — Arkansas Urology, Staff Physician

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Cooper TE, Teng C, Howell M, Teixeira-Pinto A, Jaure A, Wong G. D-mannose for preventing and treating urinary tract infections. Cochrane Database Syst Rev. 2022 Aug 30;8(8):CD013608. doi: 10.1002/14651858.CD013608.pub2. PMID 36041061